CLINICAL TRIAL: NCT00816751
Title: Paracervical Versus Intracervical Lidocaine for Suction Curettage: A Randomized Controlled Trial
Brief Title: Paracervical Versus Intracervical Lidocaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jessica Kingston, Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ONG-08-1781
Record Dates: First submitted 2008-12-31; First posted 2009-01-05 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-07

CONDITIONS: Abortion, Induced; Pain
Keywords: Local anesthesia; Paracervical; Intracervical; Abortion; Pain; Local anesthesia for elective first trimester abortion
MeSH Terms: conditions — Pain | interventions — Anesthesia, Obstetrical; Vasopressins; Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Procedure: Paracervical block; Drug: Buffered Lidocaine, vasopressin, sodium bicarbonate
- 2 (Experimental)
  Interventions: Procedure: Intracervical; Drug: Buffered Lidocaine, vasopressin, sodium bicarbonate

INTERVENTIONS:
Procedure: Paracervical block — The paracervical block was administered using 20 ml of buffered lidocaine and a 5/8 inch, 25-gauge needle. A small amount was injected at the tenaculum site, and the remainder equally distributed around the cervicovaginal junction at 3, 5, 7, and 9 o'clock. The depth was standardized at 5/8 inch by inserting the needle to the hub.
  Arms: 1
Procedure: Intracervical — The intracervical block was administered using 20 ml of buffered lidocaine and a 1-1/2 inch, 20 gauge needle in order to overcome the increased resistance to injection caused by the cervical stroma. A small amount was injected at the tenaculum site, and the remainder into the cervical stroma at 12, 3, 6, and 9 o'clock, at a depth of 1-1/2 inch by inserting the needle to the hub.
  Arms: 2
Drug: Buffered Lidocaine, vasopressin, sodium bicarbonate — The buffered lidocaine preparation for both block techniques consisted of 50 mL of 1% lidocaine, 5 units of vasopressin, and 5 mL 8% sodium bicarbonate.

SUMMARY:
The aim of this study is to estimate the efficacy of intracervical versus paracervical block on pain experienced during first trimester suction curettage without the use of preoperative cervical ripening. Because of the theoretical improved reliability of stromal block, the investigators hypothesize that intracervical block would produce lower pain scores than paracervical block at the time of cervical dilation.

ELIGIBILITY:
Inclusion Criteria:

* Women presenting for elective first trimester abortion

Exclusion Criteria:

* Gestation over 12 weeks by ultrasound
* Weight less than 98 pounds
* Known allergy to lidocaine
* Known nonviable pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2007-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Planned Parenthood, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Paracervical Block: Paracervical block: The paracervical block was administered using 20 ml of buffered lidocaine and a 5/8 inch, 25-gauge needle. A small amount was injected at the tenaculum site, and the remainder equally distributed around the cervicovaginal junction at 3, 5, 7, and 9 o'clock. The depth was standardized at 5/8 inch by inserting the needle to the hub.
  Buffered Lidocaine, vasopressin, sodium bicarbonate: The buffered lidocaine preparation for both block techniques consisted of 50 mL of 1% lidocaine, 5 units of vasopressin, and 5 mL 8% sodium bicarbonate.
- Intracervical Block: Intracervical: The intracervical block was administered using 20 ml of buffered lidocaine and a 1-1/2 inch, 20 gauge needle in order to overcome the increased resistance to injection caused by the cervical stroma. A small amount was injected at the tenaculum site, and the remainder into the cervical stroma at 12, 3, 6, and 9 o'clock, at a depth of 1-1/2 inch by inserting the needle to the hub.
  Buffered Lidocaine, vasopressin, sodium bicarbonate: The buffered lidocaine preparation for both block techniques consisted of 50 mL of 1% lidocaine, 5 units of vasopressin, and 5 mL 8% sodium bicarbonate.
Period: Overall Study
Arm/Group | Paracervical Block | Intracervical Block
Started | 45 | 44
Completed | 45 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Paracervical Block; Intracervical Block: All patients who met inclusion criteria were approached for the study. Exclusion criteria included gestational age greater than 12 weeks, patient age less than 18, patient weight less than 44 kg, patient allergy to any component of the local anesthetic, patient need for general anesthesia, inability to understand the consent form, nonviable pregnancy, current incarceration.
- Total: Total of all reporting groups
Arm/Group | Paracervical Block | Intracervical Block | Total
Number analyzed (Participants) | 45 | 44 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 44 | 89
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 44 | 89
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pain Score, as Assessed Using a 10 cm Linear Visual Analog Scale (VAS)
Description: VAS on a scale of 1 to 10 with 1 being lowest pain and 10 highest amount of pain
Time Frame: at completion of procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paracervical Block | Intracervical Block
Number analyzed (Participants) | 45 | 44
units on a scale | 4.25 (0.6) | 3.97 (0.5)

2. Secondary Outcome: Gestational Age at Time of Procedure
Time Frame: At the time of the procedure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Paracervical Block | Intracervical Block
Number analyzed (Participants) | 45 | 44
Days | 51 (11) | 54 (9)

ADVERSE EVENTS:
Arm/Group | Paracervical Block | Intracervical Block
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/44
Other Adverse Events (participants affected / at risk) | 0/45 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes